CLINICAL TRIAL: NCT05392322
Title: Effects of Virtual Video Reality Gaming on Fine Motor Skills in Children With Down's Syndrome
Brief Title: Effect of Virtual Video Reality Gaming on Fine Motor Skills in Children With Down's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0702
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Down's Syndrome; Fine Motor Skills
Keywords: Fine motor skills; Down's Syndrome; Self- help skills; Computer game
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help skills (Active Comparator): Effect of self-help skills on fine motor skills in children with down's syndrome
  Interventions: Other: Self-help skills
- Virtual video reality gaming (Experimental): Effects of virtual video reality gaming on fine motor skills in children with down's syndrome
  Interventions: Device: Virtual video reality gaming

INTERVENTIONS:
Other: Self-help skills — Self-help skills were given to down's syndrome children 3 times per week upto 15 minutes.
  Arms: Self-help skills
Device: Virtual video reality gaming — Virtual video reality gaming was given to children with down's Syndrome 3 time per week upto 15 minutes.
  Arms: Virtual video reality gaming

SUMMARY:
Down's syndrome is genetic disorder caused by trisomy 21. Children with Down's syndrome are characterized by awkward movements, gait, increased flexibility of joints, timing of mastering of basic skills, under development of fine motor skills.

Virtual Reality Therapy (VRT) is a technique that uses interactive games as a physical therapy resource and has shown positive results in cortical reorganization, improving functional mobility, and quality of movement.

This is an experimental study in which randomized controlled trials study design is being used.

DETAILED DESCRIPTION:
Down's syndrome is a genetic disorder caused by trisomy 21. Down's syndrome is characterized by a variety of dysmorphic features, congenital malformations and other health problems and medical conditions. Not all of them are present in each affected individual. The impact of Down's syndrome for each person is variable some are more affected, some are mild affected and some are fully independent.Children with Down's syndrome are characterized by awkward movements, gait, increased flexibility of joints, timing of mastering of basic skills, under development of fine motor skills.

Virtual video gaming is a best method for development of fine motor skills in Down's syndrome children. Virtual Reality Therapy (VRT) is a technique that uses interactive games as a physical therapy resource and has shown positive results in cortical reorganization, improving functional mobility, and quality of movement.

This is an experimental study in which randomized controlled trials study design is being used. Data will be collected from rising sun institute within 6 months after the approval of synopsis. Randomized sampling method will be used. Sample size will be 16 children with Down's syndrome. One group is Control group (self-help skills) in which only self-help skills effect on fine motor skills in Down's syndrome children will be assessed. Other group is Experimental group (virtual video gaming) in which effect of virtual video gaming on fine motor skills will be assessed. ABILHAND-KIDS tool will be used for measurement of effectiveness of virtual video gaming in children with Down' s syndrome. The objective of study is to determine the effects of virtual reality video gaming on fine motor skills in children with Down' s syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age group of patients ranged between 6 years to 10years.
* Both the gender will be considered.
* Subject who is able to follow the instruct

Exclusion Criteria:

* Patients with medical co-morbid.
* Gross deformity of upper /lower limb
* Epilepsy

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The abilhand-kids tool | 4th day
  The ABILHAND-KIDS tool was developed as a measure of manual ability of children with cerebral palsy. It describes most representative inventory of manual activities. The 21 items of ABILHAND-KIDS defined a valid and reliable manual ability scale. The ABILHAND-KIDS was originally developed by using the Rasch measurement model. It allows to convert ordinal score into linear measure located on unidimensional score.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, MSPPT, Principal Investigator — Riphah International University
Locations (1):
- Rising sun school for special children, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boato E, Melo G, Filho M, Moresi E, Lourenco C, Tristao R. The Use of Virtual and Computational Technologies in the Psychomotor and Cognitive Development of Children with Down Syndrome: A Systematic Literature Review. Int J Environ Res Public Health. 2022 Mar 3;19(5):2955. doi: 10.3390/ijerph19052955. PMID 35270648
- [Background] Hocking DR, Ardalan A, Abu-Rayya HM, Farhat H, Andoni A, Lenroot R, Kachnowski S. Feasibility of a virtual reality-based exercise intervention and low-cost motion tracking method for estimation of motor proficiency in youth with autism spectrum disorder. J Neuroeng Rehabil. 2022 Jan 7;19(1):1. doi: 10.1186/s12984-021-00978-1. PMID 34996473
- [Background] Klotzbier TJ, Holfelder B, Schott N. Associations of Motor Performance and Executive Functions: Comparing Children with Down Syndrome to Chronological and Mental Age-Matched Controls. Children (Basel). 2022 Jan 5;9(1):73. doi: 10.3390/children9010073. PMID 35053698
- [Background] Jain PD, Nayak A, Karnad SD, Doctor KN. Gross motor dysfunction and balance impairments in children and adolescents with Down syndrome: a systematic review. Clin Exp Pediatr. 2022 Mar;65(3):142-149. doi: 10.3345/cep.2021.00479. Epub 2021 Jun 11. PMID 34126707
- [Background] Beqaj S, Tershnjaku EET, Qorolli M, Zivkovic V. Contribution of Physical and Motor Characteristics to Functional Performance in Children and Adolescents with Down Syndrome: A Preliminary Study. Med Sci Monit Basic Res. 2018 Oct 16;24:159-167. doi: 10.12659/MSMBR.910448. PMID 30323163
- [Background] Silva V, Campos C, Sa A, Cavadas M, Pinto J, Simoes P, Machado S, Murillo-Rodriguez E, Barbosa-Rocha N. Wii-based exercise program to improve physical fitness, motor proficiency and functional mobility in adults with Down syndrome. J Intellect Disabil Res. 2017 Aug;61(8):755-765. doi: 10.1111/jir.12384. Epub 2017 Jun 6. PMID 28585394